CLINICAL TRIAL: NCT01616069
Title: Assessment and Hemodynamic Response in CABG After Cardiopulmonary Bypass Using Intraoperative Transesophegeal Echocardiography
Brief Title: Assessment of Hemodynamic Response in Cardiopulmonary Bypass Graft After Cardiopulmonary Bypass Using Transesophegeal Echocardiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other); National Institute of Cardiology/Ministry of Health (Unknown)
Responsible Party: Principal Investigator, Marcello F Salgado Filho, MD, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0362/14-12-2011
Record Dates: First submitted 2012-04-25; First posted 2012-06-11 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Cardiopulmonary Bypass Graft
Keywords: CABG; Echocardiography; Heart Failure; Heart Function
MeSH Terms: conditions — Heart Failure | interventions — Epinephrine; Simendan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epinephrine (Active Comparator): Assessment of systolic and diastolic heart function during CABAG with CPB with levosimendan using TEE.
  Interventions: Drug: epinephrine and levosimendan
- levosimendan (Active Comparator): Assessment of systolic and diastolic heart function during CABAG with CPB with epinephrine using TEE.
  Interventions: Drug: epinephrine and levosimendan

INTERVENTIONS:
Drug: epinephrine and levosimendan — epinephrine (0,06mcg/kg/min), levosimendan (0,2 mcg/kg/min)

SUMMARY:
This is a double blind randomization study, assessing hemodynamic response in patients who underwent a cardiopulmonary bypass graft (CABG) with cardiopulmonary bypass (CPB) using intraoperative trasnesophageal echocardiography (TEE) to know what inotropic drug will be batter to improve the heart function. Epinephrine, milrinone, dobutamine and levosimendan will be assessment.

ELIGIBILITY:
Inclusion Criteria:

* Sinusal ritmus
* EF > 35%
* Elective CABG surgery

Exclusion Criteria:

* No accept
* Severe valvular regurgitation or stenoses
* Chest pain
* Cardiogenic shock

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic heart function | Two years
  Assessment the systolic and diastolic heart function

SECONDARY OUTCOMES:
Mortality after CABAG | Two years
  Assessment mortality after CABAG

CONTACTS AND LOCATIONS:
Overall Officials: Marcello F Salgado Filho, Master, Principal Investigator — National Institute of Cardiology/Ministry of Health
Locations (1):
- National Institute of Cardiology / Ministry of Health, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Chung PC, Huang PC, Liu YF, Chen KB. Transesophageal echocardiography, more than a diagnostic tool: use during surgical ligation of coronary artery fistulae - a case report. J Cardiothorac Surg. 2012 Apr 6;7:28. doi: 10.1186/1749-8090-7-28. PMID 22480207
- [Result] De Mey N, Couture P, Laflamme M, Denault AY, Perrault LP, Deschamps A, Rochon AG. Intraoperative changes in regional wall motion: can postoperative coronary artery bypass graft failure be predicted? J Cardiothorac Vasc Anesth. 2012 Jun;26(3):371-5. doi: 10.1053/j.jvca.2012.02.005. Epub 2012 Mar 28. PMID 22459932
- [Result] Salgado Filho MF, Siciliano A, Siciliano A, Oliveira AJ, Salgado J, Palitot I. The importance of transesophageal echocardiography in heart harvesting for cardiac transplantation. Rev Bras Anestesiol. 2012 Mar-Apr;62(2):262-8. doi: 10.1016/S0034-7094(12)70124-1. PMID 22440381
- [Result] Fattouch K, Castrovinci S, Murana G, Novo G, Caccamo G, Bertolino EC, Sampognaro R, Novo S, Ruvolo G, Lancellotti P. Multiplane two-dimensional versus real time three-dimensional transesophageal echocardiography in ischemic mitral regurgitation. Echocardiography. 2011 Nov;28(10):1125-32. doi: 10.1111/j.1540-8175.2011.01528.x. Epub 2011 Oct 17. PMID 22004267
- [Derived] Salgado Filho MF, Barral M, Barrucand L, Cavalcanti IL, Vercosa N. A Randomized Blinded Study of the Left Ventricular Myocardial Performance Index Comparing Epinephrine to Levosimendan following Cardiopulmonary Bypass. PLoS One. 2015 Dec 14;10(12):e0143315. doi: 10.1371/journal.pone.0143315. eCollection 2015. PMID 26655803
- See also: Related Info — http://www.sba.com.br
- See also: Related Info — http://www.scahq.org